CLINICAL TRIAL: NCT06972303
Title: A Pilot Feasibility and Acceptability RCT of an App-Based Mindfulness Meditation Intervention for Sleep Among Patients With Insomnia Disorder
Brief Title: Mindfulness Meditation for Insomnia
Status: Recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Brigham and Women's Hospital (Other)
Collaborators: National Center for Complementary and Integrative Health (NCCIH) (NIH)
Responsible Party: Principal Investigator, Yan Ma, MD, MPH, Instructor, Brigham and Women's Hospital
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 2025P001314; 1K23AT012475 (NIH)
Record Dates: First submitted 2025-04-29; First posted 2025-05-15 (Actual); Last update posted 2025-12-11 (Actual); Status verified 2025-12

CONDITIONS: Sleep Initiation and Maintenance Disorders; Insomnia; Insomnia Chronic; Mindfulness; Telemedicine
MeSH Terms: conditions — Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Instructed bedtime app-guided mindfulness meditation (Experimental): Participants will utilize the specific sleep program available within the app, which will include a choice of audio soundtracks for guided MM (no exposure to screen lights during practice). The practice may involve techniques such as breathing exercise, imagery, body scan, and relaxation. Participants will specifically use the app during the immediate pre-sleep period. They can choose their preferred meditation sessions within the Sleep menu in Week 1-4.
  Interventions: Behavioral: Instructed bedtime app-guided mindfulness meditation; Behavioral: Sleep hygiene education
- Uninstructed app-guided mindfulness meditation (Experimental): Participants will be asked to practice MM using the same app during daytime (prior to the evening meal), but without specific study instructions around components to access or specific time of practice.
  Interventions: Behavioral: Uninstructed app-guided mindfulness meditation; Behavioral: Sleep hygiene education
- Sleep Hygiene Education only (Other): Participants will receive sleep hygiene education and asked not to start any new insomnia treatments. Sleep hygiene education serves as a minimal intervention control condition and real-world comparator. At the end of the study, interested participants in the control group will be given equal access to the mobile app. Usual care for insomnia typically involves sleep hygiene education, so all three groups will receive standard SHE as part of usual care.
  Interventions: Behavioral: Sleep hygiene education

INTERVENTIONS:
Behavioral: Instructed bedtime app-guided mindfulness meditation — All participants will access the a smartphone app, and the mindfulness meditation practice may involve techniques such as breathing exercise, imagery, body scan, and relaxation. The investigators will provide instructions for participants who are assigned to practice at bedtime.
  Other Names: Uninstructed bedtime app-guided mindfulness meditation; Sleep hygiene education
  Arms: Instructed bedtime app-guided mindfulness meditation
Behavioral: Uninstructed app-guided mindfulness meditation — The guided mindfulness meditation practice will also be based on the same app. The investigators will not provide instructions for participants, and they have complete freedom to use the app as real-world users.
  Arms: Uninstructed app-guided mindfulness meditation
Behavioral: Sleep hygiene education — Sleep hygiene education will be based on recognized, general, non-personalized sleep hygiene advice, for example, recommendations about bedtime routines and use of alcohol and caffeine, tips on creating a sleep-conducive bedroom environment.

SUMMARY:
The investigators will conduct a 3-arm, pilot RCT where participants (N=30) will be randomized in a 1:1:1 design to 4 weeks of instructed bedtime MM practice at night (n=10) vs. uninstructed MM (n=10) vs. sleep hygiene education only (n=10). Aim 1 is to understand the feasibility and acceptability of the intervention and study procedures. Aim 2 is to explore patterns of within-group changes in sleep outcomes (i.e., insomnia severity and sleep quality). Patient-reported outcomes will be collected using a HIPAA-compliant electronic data management system (REDCap). Following informed consent, participants will receive links to REDCap surveys via email at Weeks 0, 4, 8, and 16. The investigators will also conduct a post-intervention interview at the end of Week 4 and an exit interview at Week 16. All participants will also receive a research kit with wearable devices and meet with our staff after they receive the kit for instructions. Data collected in the pilot RCT will help us to preliminarily identify tools for subjective measures and physiological signals to inform a future trial.

ELIGIBILITY:
Inclusion Criteria:

* Age 18 years and older;
* Chronic insomnia (≥ 3 nights/week, for ≥ 3 months), defined by DSM-V or ICSD-3;
* Have a primary complaint of difficulty falling asleep (sleep-onset insomnia) with self-reported sleep onset latency >20 min;
* Insomnia Severity Index score ≥ 15;
* Speak and understand English;
* Have a smart device (phone or tablet) for mobile app installation

Exclusion Criteria:

* Current diagnosis of sleep disorders other than insomnia (e.g., narcolepsy, restless leg syndrome, REM sleep behavior disorder, etc.);
* Shift worker or routine night shifts;
* Women with pregnancy or breastfeeding;
* Regular (defined as twice a week or more) practice of mind-body interventions;
* Patients with pace-maker or routinely using cardiovascular medications that have effects on heart rates (i.e., beta-blockers);
* Neurological disorders (e.g. epilepsy, dementia, stroke, Parkinson's disease, neuroinfections, brain tumors, etc.) or current diagnosis of comorbid psychotic, substance use, and trauma-related disorders;
* Currently under medications with sleep changing effects (e.g., anxiolytics/benzodiazepines, selective serotonin reuptake inhibitors, hypnotics, etc.);
* Hearing impairment or loss. Participants will be asked to report any medication for at least 2 weeks prior to study onset and during the study period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-12 (Estimated); Primary Completion 2028-07-31 (Estimated); Study Completion 2028-12-29 (Estimated)

PRIMARY OUTCOMES:
Screened-to-eligible ratio | Week 0
  The proportion of screened participants who were determined to be eligible for the study; calculated as the number of eligible participants divided by the total number of individuals screened.
Retention rate | Weeks 4, 8, and 16
  Retention rate is defined as the percentage of participants who complete the entire follow-up period. Reasons for participant dropout will also be documented.
Adherence to intervention protocol | Week 4
  In the intervention groups, a mindfulness meditation session ≥ 10 minutes will be considered as a completed session. Numbers of sessions completed during the four weeks will be recorded. Adherence to intervention protocol will be defined as those randomized to the intervention groups complete ≥ 70% of home practice.
Compliance with outcome assessment | Weeks 0, 4, 8, 16
  Compliance with outcome assessment will be determined by the percentage of participants who complete ≥ 70% of questionnaires at each time point.
Acceptability | Week 4
  At intervention end (week 4), a brief questionnaire will ask participants to rate (1=not at all to 5=very much) the enjoyableness, convenience, helpfulness, and overall satisfaction with the app-based mindfulness practice. Acceptability is assessed by self-report survey ratings, and a threshold of 80% ratings of 4 or higher will indicate acceptability.

SECONDARY OUTCOMES:
Insomnia severity | Weeks 0, 4, 8, 16
  Insomnia severity will be assessed by the Insomnia Severity Index (ISI), a brief instrument that assesses insomnia. Its reliability, validity, and sensitivity to treatment response have been documented in the general population and with patients with insomnia. The total score ranges from 0 to 28, and higher scores indicate more severe insomnia. This secondary/exploratory outcome will be summarized with simple descriptive statistics without formal efficacy testing.
Sleep quality | Weeks 0, 4, 8, 16
  Sleep quality will be assessed by the Pittsburgh Sleep Quality Index (PSQI). PSQI is a subjective sleep assessment, which includes multiple sleep-related variables over the preceding month. The PSQI yields seven component scores: subjective sleep quality, sleep latency, sleep duration, habitual sleep efficiency, sleep disturbances, sleep medication, and daytime dysfunction. The global score ranges from 0 to 21, and higher scores suggest greater sleep disturbance. This secondary/exploratory outcome will be summarized with simple descriptive statistics without formal efficacy testing.

CONTACTS AND LOCATIONS:
Locations (1):
- Brigham and Women's Hospital, Boston, Massachusetts, United States